CLINICAL TRIAL: NCT00192075
Title: A Multicenter, Randomized Phase II Trial of Avastin Plus Gemcitabine Plus 5FU/Folinic Acid (A + FFG) vs. Avastin Plus Oxaliplatin Plus 5FU/Folinic Acid (A + FOLFOX 4) as Therapy for Patients With Metastatic Colorectal Cancer
Brief Title: A Randomized Trial of Avastin + Gemcitabine + 5-Fluorouracil (5FU)/Folinic Acid Versus Avastin + Oxaliplatin + 5FU/Folinic Acid in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly and Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8142; B9E-US-S337 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2009-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gemcitabine; Bevacizumab; Oxaliplatin

ARMS (2):
- A+FFG (Experimental): Avastin + Gemcitabine + 5-Fluorouracil (5FU)/Folinic Acid
  Interventions: Drug: Gemcitabine; Drug: avastin; Drug: 5FU/folinic acid
- A+FOLFOX 4 (Active Comparator): Avastin + Oxaliplatin + 5-Fluorouracil (5FU)/Folinic Acid
  Interventions: Drug: avastin; Drug: 5FU/folinic acid; Drug: oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — 900 mg/m2 IV over 90 minutes after Folinic Acid weekly for 6 weeks every 8 weeks until progression.
  Other Names: Gemzar
  Arms: A+FFG
Drug: avastin — 5 milligrams per kilogram (mg/kg)
Drug: 5FU/folinic acid — Folinic Acid: 100 milligrams per square meter (mg/m2) intravenous (IV) over 60 minutes (A+FFG).
  Folinic Acid: 200 mg/m2 as a 2-hr infusion on Days 1 and 2 of a 14-day cycle (A+FOLFOX 4).
  5-Fluorouracil: 450 mg/m2 as an IV bolus in middle of Folinic Acid (A+FFG). 5-Fluorouracil: 400 mg/m2 bolus plus a 600 mg/m2 22-hour infusion on Days 1 and 2 of a 14-day cycle (A+FOLFOX 4).
Drug: oxaliplatin — 85 mg/m2 as a 2-hour infusion on Day 1 of a 14 day cycle.
  Arms: A+FOLFOX 4

SUMMARY:
The purpose of the study is to describe the tumor response rates for the two regimens being studied, and to determine how long patients live after receiving the treatment, how long patients are without return of their disease after they receive treatment, and how long the response they get from the treatment lasts. The amount and type of side effects/toxicities of each regimen will also be evaluated. The regimen including Oxaliplatin + 5FU/Folinic Acid is a current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or cytological diagnosis of the colon or rectum with Stage III unresectable or Stage IV disease.
* Urinalysis or Urine dipstick for proteinuria of less than 1+ (i.e. either 0 or trace). If urine dipstick is greater than 1+, the 24 hour urine protein must demonstrate less than 500 mg of protein in 24 hours to allow participation.
* No prior chemotherapy, immunotherapy, or hormonal treatment for metastatic disease is acceptable. However, one prior neo-adjuvant or adjuvant treatment is acceptable, including Capecitabine, Camptothecin-11 (CPT-11), 5 Fluorouracil/Leucovorin (5FU/LV) or Radiation containing regimens, (but no Oxaliplatin), and only if progression > 6 months since last adjuvant treatment.
* Prior radiation therapy, including radiation to the whole pelvis, is allowed (Cristy and Eckerman 1987) and patients must have recovered from the acute toxic effects of the treatment prior to study enrollment. Prior palliative radiation therapy given to a non-measurable diagnostic site is acceptable if given > 4 weeks prior to treatment or if other non-irradiated measurable disease is present.
* No known central nervous system (CNS) metastasis.

Exclusion Criteria:

* Histology other than adenocarcinoma
* Tumors that demonstrate free perforation as manifested by free air or free fluid in the abdomen. Patients with walled-off perforation are eligible.
* Gastroduodenal ulcer determined as active by endoscopy.
* Invasive procedures defined as follows; major surgical procedures, open biopsy, or significant traumatic injury within 28 days prior to randomization, anticipation of need for major surgical procedure during the course of study, core biopsy or other minor procedure within 7 days prior to registration.
* Following cardiac condition; New York Heart Association (NYHA) Class III or IV, myocardial infarction (MI) within 6 months, unstable angina within 6 months and current symptomatic arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-06; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tupelo, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin

REFERENCES:
- [Result] Madajewicz S, Waterhouse DM, Ritch PS, Khan MQ, Higby DJ, Leichman CG, Malik SK, Hentschel P, Gill JF, Zhao L, Nicol SJ. Multicenter, randomized phase II trial of bevacizumab plus folinic acid, fluorouracil, gemcitabine (FFG) versus bevacizumab plus folinic acid, fluorouracil, oxaliplatin (FOLFOX4) as first-line therapy for patients with advanced colorectal cancer. Invest New Drugs. 2012 Apr;30(2):772-8. doi: 10.1007/s10637-010-9598-9. Epub 2010 Dec 1. PMID 21120580

RESULTS

PARTICIPANT FLOW:
Groups:
- A+FFG: Includes all patients in the intent-to-treat population including patients administered Avastin (Avastin plus gemcitabine plus 5FU/Folinic Acid)
- A + FOLFOX 4: Includes all patients in the intent-to-treat population including patients administered Avastin (Avastin plus oxaliplatin plus 5FU/Folinic Acid)
Period: Overall Study
Arm/Group | A+FFG | A + FOLFOX 4
Started | 42 | 42
Completed | 3 | 23
Not Completed | 39 | 19
Not completed — Disease Progression | 23 | 6
Not completed — Adverse Event | 1 | 3
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Patient Non-Compliance | 0 | 1
Not completed — Unacceptable Toxicity Exhibited by Drug | 2 | 1
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A+FFG | A + FOLFOX 4 | Total
Number analyzed (Participants) | 42 | 42 | 84
Age Continuous [Median (Full Range); unit: years] | 62 [28 to 79] | 64 [32 to 81] | 63 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 21 | 20 | 41
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84
Diagnosis to Enrollment [Number; unit: participants]
  <6 months | 29 | 29 | 58
  >=6 months | 13 | 13 | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 23 | 20 | 43
    1 - Ambulatory, Restricted Strenuous Activity | 19 | 22 | 41
Primary Tumor Site [Number; unit: participants]
  Colon | 25 | 35 | 60
  Rectum | 10 | 4 | 14
  Other | 7 | 3 | 10
Prior Adjuvant Therapy [Number; unit: participants]
  Yes | 12 | 14 | 26
  No | 30 | 28 | 58
Race/Ethnicity [Number; unit: participants]
  Caucasian | 33 | 34 | 67
  African descent | 5 | 6 | 11
  Asian | 0 | 1 | 1
  Hispanic | 4 | 1 | 5
Site of Metastasis [Number; unit: participants] — Metastasis could occur in multiple sites.
  participants
    Liver | 28 | 29 | 57
    Lung | 13 | 11 | 24
    Abdominal | 3 | 3 | 6
    Regional lymph nodes | 14 | 14 | 28
    Distant lymph nodes | 4 | 3 | 7
    Genitourinary | 1 | 0 | 1
    Other | 8 | 3 | 11
Tumor Stage [Number; unit: participants] — Patients could experience multiple tumors.
  participants
    Primary tumor | 37 | 41 | 78
    Regional lymph nodes | 24 | 29 | 53
    Distant metastasis | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response by Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | A+FFG | A + FOLFOX 4
Number analyzed (Participants) | 42 | 42
participants
  Complete Response (CR) | 1 | 2
  Partial Response (PR) | 3 | 15
  Overall Response Rate (CR+PR) | 4 | 17
  Stable Disease (SD) | 21 | 16
  Disease Control Rate (CR+PR+SD) | 25 | 33
  Progressive Disease | 14 | 7
  Unknown | 3 | 2

2. Secondary Outcome: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: randomization to the date of first documented disease progression or death due to disease under study, whichever comes first (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: Intent to treat population. Five patients in A+FFG and 5 patients in A+FOLFOX4 were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+FFG | A + FOLFOX 4
Number analyzed (Participants) | 42 | 42
months | 8.6 [5.3 to 17.9] | 9.7 [7.3 to 11.2]

3. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from randomization to the first observation of disease progression, or death due to any cause.
Time Frame: randomization to the first date of progression or death from any cause (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: Intent to treat population. Three patients in A+FFG and 4 patients in A+FOLFOX4 were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+FFG | A + FOLFOX 4
Number analyzed (Participants) | 42 | 42
months | 8.6 [4.7 to 17.9] | 9.5 [6.9 to 11.2]

4. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: randomization to the date of death from any cause (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: Intent to treat population. Eight patients in A+FFG and 12 patients in A+FOLFOX4 were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+FFG | A + FOLFOX 4
Number analyzed (Participants) | 42 | 42
months | 20.6 [14.8 to 26.7] | 19.7 [11.2 to 32.0]

5. Other Pre Specified Outcome: Tumor Response - Avastin Subgroup
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The original treatment regimens were FFG and FOLFOX. Due to FDA approval of Avastin, protocol was amended to add Avastin to treatment regimens. This is the population of patients who received Avastin with the original treatment.
Measure: Number; unit: participants
Groups:
- A+FFG - Avastin Subgroup: Patients who received Avastin plus gemcitabine plus 5FU/Folinic Acid
- A + FOLFOX 4 - Avastin Subgroup: Patients who received Avastin plus oxaliplatin plus 5FU/Folinic Acid
Arm/Group | A+FFG - Avastin Subgroup | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 18 | 18
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 0 | 8
  Overall Response Rate (CR+PR) | 0 | 9
  Stable Disease (SD) | 11 | 8
  Disease Control Rate (CR+PR+SD) | 11 | 17
  Progressive Disease | 6 | 1
  Unknown | 1 | 0

6. Other Pre Specified Outcome: Time to Progressive Disease - Avastin Subgroup
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The original treatment regimens were FFG and FOLFOX. Due to FDA approval of Avastin, protocol was amended to add Avastin to treatment regimens. This is the population of patients who received Avastin with the original treatment. Three patients in A+FFG - Avastin subgroup and 4 patients in A+FOLFOX4 - Avastin subgroup were censored.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- A + FOLFOX 4 - Avastin Subgroup: Includes patients who received Avastin plus oxaliplatin plus 5FU/Folinic Acid
Arm/Group | A+FFG - Avastin Subgroup | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 18 | 18
months | 13.7 [4.6 to 19.3] | 13.8 [6.3 to 23.7]

7. Other Pre Specified Outcome: Progression-Free Survival - Avastin Subgroup
Description: Defined as the time from date of first dose to the first observation of disease progression, or death due to any cause.
Time Frame: as for outcome 3
Population: The original treatment regimens were FFG and FOLFOX. Due to FDA approval of Avastin, protocol was amended to add Avastin to treatment regimens. This is the population of patients who received Avastin with the original treatment. Three patients in A+FFG - Avastin subgroup and 3 patients in A+FOLFOX4 - Avastin subgroup were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+FFG - Avastin Subgroup | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 18 | 18
months | 13.7 [4.6 to 19.3] | 11.5 [6.3 to 18.1]

8. Other Pre Specified Outcome: Survival at 12 Months and 24 Months - Avastin Subgroup
Description: Percentage of participants who were alive at 12 months and 24 months.
Time Frame: randomization to the date of death from any cause (up to 24 months)
Population: The original treatment regimens were FFG (Arm A) and FOLFOX (Arm B). Due to FDA approval of Avastin, protocol was amended to add Avastin to treatment regimens. This is the population of patients who received Avastin with the original treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants alive
Arm/Group | A+FFG - Avastin Subgroup | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 18 | 18
percentage of participants alive
  12-Month Survival | 75.6 [47.3 to 90.1] | 83.3 [56.8 to 94.3]
  24-Month Survival | 50.4 [24.9 to 71.4] | 66.7 [40.4 to 83.4]

9. Other Pre Specified Outcome: Toxicity - Avastin Subgroup
Description: Includes all Grade 3-4 hematologic toxicities and all non-hematologic toxicities with either >=1 Grade 4 or >=2 Grade 3 adverse events
Time Frame: every cycle (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- A+FFG - Avastin Subgrouup: Patients who received Avastin plus gemcitabine plus 5FU/Folinic Acid
Arm/Group | A+FFG - Avastin Subgrouup | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 18 | 18
participants
  Neutropenia (Grade 3) | 3 | 5
  Neutropenia (Grade 4) | 5 | 1
  Thrombocytopenia (Grade 3) | 1 | 0
  Thrombocytopenia (Grade 4) | 0 | 0
  Leukopenia (Grade 3) | 3 | 0
  Leukopenia (Grade 4) | 1 | 0
  Anemia (Grade 3) | 0 | 0
  Anemia (Grade 4) | 0 | 0
  Febrile neutropenia (Grade 3) | 0 | 1
  Febrile neutropenia (Grade 4) | 0 | 0
  Diarrhea (Grade 3) | 1 | 0
  Diarrhea (Grade 4) | 0 | 1
  Small intestinal obstruction (Grade 3) | 1 | 1
  Small intestinal obstruction (Grade 4) | 0 | 0
  Fatigue (Grade 3) | 0 | 2
  Fatigue (Grade 4) | 0 | 0
  Cerebral infarction (Grade 3) | 0 | 0
  Cerebral infarction (Grade 4) | 0 | 0
  Hyperglycemia (Grade 3) | 0 | 0
  Hyperglycemia (Grade 4) | 0 | 0
  Dehydration (Grade 3) | 0 | 1
  Dehydration (Grade 4) | 0 | 0
  Deep vein thrombosis (Grade 3) | 0 | 2
  Deep vein thrombosis (Grade 4) | 0 | 0
  Myocardial infarction (Grade 3) | 0 | 0
  Myocardial infarction (Grade 4) | 0 | 2
  Subdural hematoma (Grade 3) | 0 | 0
  Subdural hematoma (Grade 4) | 0 | 0
  Perirectal abscess (Grade 3) | 1 | 0
  Perirectal abscess (Grade 4) | 0 | 0
  Hypoxia (Grade 3) | 0 | 0
  Hypoxia (Grade 4) | 0 | 0

10. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: date of first response until the first date of documented progression or death from any cause (every 7-8 weeks for 2 cycles, monthly for 3 months, every other month for 6 months, then every 3 months up to 4.4 years)
Population: Intent to treat population who were responders (had best overall response of either complete response or partial response). Zero patients in A+FFG and 2 patients in A+FOLFOX4 were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+FFG | A + FOLFOX 4
Number analyzed (Participants) | 4 | 17
months | 12.7 [5.5 to 32.9] | 7.9 [4.4 to 9.8]

11. Other Pre Specified Outcome: Duration of Response - A+FOLFOX4 - Avastin Subgroup
Description: as for outcome 10
Time Frame: as for outcome 10
Population: The original treatment regimens were FFG and FOLFOX. Due to FDA approval of Avastin, protocol was amended to add Avastin to treatment regimens. This is the population of patients who received Avastin with the original treatment. Results were not calculable for the A+FFG-Avastin subgroup. Two patients were censored in the A+FOLFOX4-Avastin subgroup.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- A + FOLFOX 4 - Avastin Subgroup: Includes all patients in the intent-to-treat population including patients administered Avastin (Avastin plus oxaliplatin plus 5FU/Folinic Acid)
Arm/Group | A + FOLFOX 4 - Avastin Subgroup
Number analyzed (Participants) | 9
months | 5.2 [4.2 to 13.8]

ADVERSE EVENTS:
Arm/Group | A+FFG | A + FOLFOX 4
Serious Adverse Events (participants affected / at risk) | 11/42 | 8/42
Other Adverse Events (participants affected / at risk) | 40/42 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A+FFG (N=42) | A + FOLFOX 4 (N=42)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perirectal abscess (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A+FFG (N=42) | A + FOLFOX 4 (N=42)
Anaemia (Blood and lymphatic system disorders) | 16 (32) | 4 (6)
Leukopenia (Blood and lymphatic system disorders) | 8 (29) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 24 (76) | 16 (34)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (37) | 8 (13)
Abdominal pain (Gastrointestinal disorders) | 9 (15) | 4 (5)
Constipation (Gastrointestinal disorders) | 15 (39) | 10 (16)
Diarrhoea (Gastrointestinal disorders) | 15 (30) | 17 (38)
Dry mouth (Gastrointestinal disorders) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (39) | 25 (49)
Stomatitis (Gastrointestinal disorders) | 9 (14) | 5 (5)
Vomiting (Gastrointestinal disorders) | 8 (18) | 15 (26)
Asthenia (General disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 22 (46) | 24 (48)
Oedema peripheral (General disorders) | 3 (5) | 4 (4)
Pain (General disorders) | 3 (4) | 3 (4)
Pyrexia (General disorders) | 10 (16) | 6 (6)
Rigors (General disorders) | 6 (9) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Haematocrit decreased (Investigations) | 5 (7) | 2 (4)
Haemoglobin decreased (Investigations) | 6 (9) | 4 (13)
Neutrophil count decreased (Investigations) | 8 (20) | 7 (14)
Neutrophil percentage decreased (Investigations) | 3 (5) | 2 (7)
Platelet count decreased (Investigations) | 5 (7) | 5 (7)
Red blood cell count decreased (Investigations) | 3 (3) | 1 (2)
Weight decreased (Investigations) | 5 (5) | 1 (1)
White blood cell count decreased (Investigations) | 8 (18) | 5 (7)
White blood cell count increased (Investigations) | 0 (0) | 3 (10)
Anorexia (Metabolism and nutrition disorders) | 8 (16) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (14) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Dysgeusia (Nervous system disorders) | 5 (5) | 6 (7)
Headache (Nervous system disorders) | 10 (21) | 3 (4)
Neuropathy (Nervous system disorders) | 0 (0) | 9 (13)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 7 (9)
Paraesthesia (Nervous system disorders) | 2 (2) | 11 (25)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 6 (21)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (5) | 3 (3)
Proteinuria (Renal and urinary disorders) | 5 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 6 (7)
Flushing (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days